CLINICAL TRIAL: NCT00640120
Title: Wheeze Detection in Children During Dynamic Bronchial Situations Measured by WIM-PC™ Recording
Status: Completed | Type: Observational
Sponsor: KarmelSonix Ltd. (Industry)
Responsible Party: Dr. Hanna Levy, KarmelSonix Ltd
Other Study IDs: KSI-WZK-01
Record Dates: First submitted 2008-03-15; First posted 2008-03-21 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2008-03

CONDITIONS: Asthma, Bronchial
Keywords: wheeze detection
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Asthmatic subjects
  Interventions: Device: WIM-PC™ device
- 2: Healthy subjects
  Interventions: Device: WIM-PC™ device

INTERVENTIONS:
Device: WIM-PC™ device — wheeze detection during dynamic bronchial situations in infants

SUMMARY:
The WIM-PC™ device, indicated for acoustic pulmonary function measurement that quantifies the presence of wheezing. This study was designed in order to evaluate the efficacy and safety of using the WIM-PC™ device for wheeze detection during dynamic bronchial situations in infants that were hospitalized as a result of asthmatic attack.

DETAILED DESCRIPTION:
Asthma is the most common cause of hospitalization for respiratory infection in infants under one year of age. About 1-2% of infants with bronchiolitis need to be hospitalized and approximately 8% of these children require intensive care. Pulmonary function tests in infants are objective, but require sedation, which is problematic in acutely ill infants. Wheeze quantification by lung sounds analysis methods is objective, non invasive and has been shown to correlate with clinical status in asthma and bronchiolitis. The recording procedure is simple, requiring only the attachment of 4 ECG-size sensors to the chest wall. A 30-second recording is often adequate, but recording time can be extended as necessary, to obtain good quality data, where wheezes are detected and counted with high degree of accuracy.

Karmel Sonix Ltd has developed the WIM-PC™ device, indicated for acoustic pulmonary function measurement that quantifies the presence of wheezing. This study was designed in order to evaluate the efficacy and safety of using the WIM-PC™ device for wheeze detection during dynamic bronchial situations in infants that were hospitalized as a result of asthmatic attack.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic or healthy subjects;
* Age up to 18 years;
* Subject or subject's parents/guardian is able to comprehend and give informed consent for participation in the study.

Exclusion Criteria:

* Chest lesions (rush or deformity);
* Hemodynamic instability;
* Concurrent additional major illness.
* Concurrent participation in any other clinical study.
* Physician objection.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: asthmatic subjects or healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Study success will be declared if one of the following is met: A correlation of at least 0.25 (R2=0.25) will be found between WR and FEV1 measurements; A correlation of at least 0.7 will be found between clinical parameter and WZ measurements. | 6 months

SECONDARY OUTCOMES:
Evaluation of the safety of using the WIM-PC™ for wheeze detection. Safety will be established by lack of adverse events. Since this is a Non Significant Risk (NSR) device serious adverse events are not expected | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Noam Gavriely, Prof., Study Director
Locations (1):
- Bnei-Zion Medical Center, Haifa, Israel